CLINICAL TRIAL: NCT02809443
Title: Phase I, Open-label, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of GLS-5700 Administered ID Followed by EP in Dengue Virus-Naïve Adults
Brief Title: GLS-5700 in Dengue Virus-Naïve Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Zika-001
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Zika; Vaccine; DNA
MeSH Terms: conditions — Zika Virus Infection | interventions — GLS-5700 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLS-5700 at 1 mg (Experimental): DNA/dose
  Interventions: Biological: GLS-5700
- GLS-5700 at 2 mg (Experimental): DNA/dose
  Interventions: Biological: GLS-5700

INTERVENTIONS:
Biological: GLS-5700 — GLS-5700 contains a single plasmid containing DNA encoding for pre-membrane and envelope (prME) proteins of the Zika virus

SUMMARY:
The clinical trial will assess the safety, tolerability, and immunogenicity of GLS-5700. GLS-5700 is a synthetic DNA plasmid vaccine against the Zika virus. ZIKA-001 is the first in man clinical trial of this vaccine which encodes for the premembrane-membrane and envelope regions of Zika virus.

DETAILED DESCRIPTION:
GLS-5700 contains a single plasmid containing DNA encoding for pre-membrane and envelope (prME) proteins of the Zika virus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. Able to provide consent to participate and having signed an Informed Consent Form (ICF);
3. Able and willing to comply with all study procedures;
4. Women of child-bearing potential agree to use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile from enrollment to 3 months following the last injection, or have a partner who is medically unable to induce pregnancy.
5. Sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception during the study, and agree to continue the use for at least 3 months following the last injection, or have a partner who is permanently sterile or is medically unable to become pregnant;
6. Normal screening ECG or screening ECG with no clinically significant findings;
7. Screening laboratory must be within normal limits or have only Grade 0-1 findings;
8. No history of clinically significant immunosuppressive or autoimmune disease.
9. No history of dengue virus vaccination or illness; no history of yellow fever vaccination.
10. Dengue seronegative at baseline by screening laboratory evaluation
11. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day).

Exclusion Criteria:

1. Administration of an investigational compound either currently or within 30 days of first dose;
2. Previous receipt of an investigational product for the treatment or prevention of Zika virus except if participant is verified to have received placebo;
3. Administration of any vaccine within 4 weeks of first dose;
4. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose
5. Administration of any blood product within 3 months of first dose;
6. Pregnancy or breast feeding or plans to become pregnant during the course of the study;
7. Positive serologic result for dengue virus (any serotype) or history of receipt of either dengue virus or yellow fever virus vaccination at any time in the past;
8. Positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
9. Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
10. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 (CKD Stage II or greater);
11. Baseline screening lab(s) with Grade 2 or higher abnormality, except for Grade 2 creatinine;
12. Chronic liver disease or cirrhosis;
13. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
14. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day);
15. Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
16. Prior major surgery or any radiation therapy within 4 weeks of group assignment;
17. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
18. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD)
19. Metal implants within 20 cm of the planned site(s) of injection;
20. Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection.
21. Prisoner or participants who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
22. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
23. Not willing to allow storage and future use of samples for Zika virus related research
24. Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Maslow, MD, Study Chair — GeneOne Life Science
Locations (3):
- United States (2):
  - Miami Research Associate, Miami, Florida
  - University of Pennslyvania, Philadelphia, Pennsylvania
- CHU de Québec -Université Laval hopital CHUL Centre de Recherche en infectiologie, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tebas P, Roberts CC, Muthumani K, Reuschel EL, Kudchodkar SB, Zaidi FI, White S, Khan AS, Racine T, Choi H, Boyer J, Park YK, Trottier S, Remigio C, Krieger D, Spruill SE, Bagarazzi M, Kobinger GP, Weiner DB, Maslow JN. Safety and Immunogenicity of an Anti-Zika Virus DNA Vaccine. N Engl J Med. 2021 Sep 16;385(12):e35. doi: 10.1056/NEJMoa1708120. PMID 34525286

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg
Started | 20 | 20
Completed | 17 | 19
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.19) | 42.6 (14.25) | 41.2 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 13 | 18 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events From Day 0 Through Week 60
Time Frame: Day 0 through Week 60
Measure: Number; unit: participants
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

2. Secondary Outcome: Binding Antibody Response to Zika Envelope
Description: Serum samples were analyzed on enzyme-linked immunosorbent assay (ELISA) to measure binding-antibody responses to recombinant vaccine-matched ZIKV envelope (rZIKV-E) protein and reported as the number of participants who responded.
Time Frame: Week 14 (2 weeks after the 3rd dose)
Population: Participants who had received all 3 doses of GLS-5700 in a 1-mg or 2-mg dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg
Number analyzed (Participants) | 20 | 19
Participants | 20 | 19

3. Secondary Outcome: T Cell Response
Description: PBMCs were tested in enzyme-linked immunospot (ELISPOT) assay to detect the production of interferon-γ-secreting cells in response to stimulation with ZIKV premembrane and envelope peptides
Time Frame: Maximum response over follow up period up to 60 weeks.
Measure: Median (Inter-Quartile Range); unit: Spot Forming Units per million cells
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg
Number analyzed (Participants) | 18 | 19
Spot Forming Units per million cells | 35 [15 to 72] | 154 [42 to 283]

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from Week 0 through Week 60.
Description: Adverse events were graded according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials guidelines that were issued by the Food and Drug Administration in September 2007.
Arm/Group | GLS-5700 at 1 mg | GLS-5700 at 2 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLS-5700 at 1 mg (N=20) | GLS-5700 at 2 mg (N=20)
Pain at injection site (Surgical and medical procedures) | 20 (20) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02809443/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02809443/SAP_001.pdf